CLINICAL TRIAL: NCT04714034
Title: Real Risks of the Online World: Association of Problematic Online Dating App Use with Mental and Sexual Health Outcomes in Sexual Minorities
Brief Title: Real Risks of the Online World
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital of Psychiatry Zurich (Unknown); Center for Forensic Hair Analysis, Zurich (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-01545; 10001C_192814 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2020-12-13; First posted 2021-01-19 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Sexual Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV-negative SwissPrePared participants who are active Online Dating App (ODA) users
  Interventions: Diagnostic Test: to develop and validate a scale measuring problematic online dating app (ODA) use in sexual minorities

INTERVENTIONS:
Diagnostic Test: to develop and validate a scale measuring problematic online dating app (ODA) use in sexual minorities — Qualitative part: scale development and validation with testing in 3 different participant samples, i.e. preliminary testing (n=10), pilot testing (n=30-60), validation (n=300).
  Quantitative part: longitudinal part conducted in the validation sample of the qualitative study part (n=300) with the aim to evaluate the association of scores in the problematic ODA use scale with sexual health and mental health outcomes.

SUMMARY:
Development and validation of questionnaire/scale to assess problematic online dating app (ODA) use in a sub-cohort of the SwissPrEPared cohort study (validation sample: n=229). Longitudinal design to assess the association of problematic ODA use and sexual/mental health and substance use outcomes. No randomised trial, only 1 cohort which will be stratified according to severity/risk of problematic ODA use.

DETAILED DESCRIPTION:
This project may fill an important gap of knowledge in a research area that has taken on major importance over the past few years, and has thus the potential to impact several major public health recommendations. First, considering the high penetrance of dating apps in the men who have sex with men (MSM) population (reaching 78.2% in a recent report), more than 62,000 MSM in Switzerland are estimated to use such applications. How many of them suffer from addiction or problmatic use remains unclear and our project will be the first to provide estimates of the prevalence of problematic ODA use in this particular population. Second, our project will help to clarify the impact of online dating app usage on health outcomes. By identifying drivers of the current HIV/(sexual transmitted infections (STI) epidemic in Switzerland, our project might thus provide critical information to shape future prevention measures aiming at further reducing HIV/STI incidence rates. Third, because sexual risk-taking increases with substance use and depression, it remains crucial to detect mental health outcomes early and provide adequate care to populations at high risk of HIV, or other STI, transmission. Fourth, our study might identify a new phenomenon related to high-risk sexual behaviour that may not be limited to the MSM group, but could also affect other, larger populations interacting and meeting through online communication channels. Considering that more than 41 million people are currently using dating apps in Europe, our findings might have a substantial impact on the general population. Finally, this project might provide the very first insights on the interplay between online dating, substance use, mental health and sexual risk taking. This new understanding could then help Switzerland create additional measures for preventing HIV transmission and reach the UNAIDS targets for HIV elimination by 2030.

ELIGIBILITY:
Inclusion Criteria:

* currently engaging in online dating (i.e., using applications/websites with the aim to meet potential relationship or sexual partners or having used them actively in the past 12 months)
* Participating in the SwissPrEPared study at center Checkpoint Zurich
* German speaking

Exclusion Criteria:

- Potential participants will be excluded if they are unable to follow study procedures.

For Inclusion/Exclusion at the SwissPrEPared study see: NCT03893188 at clinicaltrials.gov

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-negative SwissPrEPared participants (≥ 18 years old) who are active online dating app users.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Develop and validate a scale measuring problematic online dating app (ODA) use | single measurement (one day per participant)
  Scale development and validation will follow the FDA guidance for patient-reported outcomes and recommendations on questionnaire research. Preliminary testing, pilot-testing, and validation will be conducted in participants from the SwissPrEPared Study
Associated mental, sexual health and substance use outcomes of problematic ODA use | 6 months
  Evaluate the association of problematic ODA use with:
  Sexual health outcomes (incident cases of STI, such as syphilis, gonorrhoea and chlamydia, or HIV), over 6 months Mental health outcomes: prevalence of psychiatric disorders, measured at baseline and 12 months, using validated questionnaires Substance use outcomes: Lifetime, 12-month, 3-month prevalence and frequency rates

CONTACTS AND LOCATIONS:
Locations (1):
- Epidemiology, Biostatistics and Prevention Institute, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No